CLINICAL TRIAL: NCT05668637
Title: Retrospective Use of Patient Treatment Data for the Evaluation and Further Development of an Artificial Intelligence-based Algorithm for Clinical Decision Support in Invasive Mechanical Ventilation of Intensive Care Patients
Brief Title: Evaluation and Further Development of an Artificial Intelligence-based Algorithm for Clinical Decision Support
Acronym: IntelliLung
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: TUD-IntelliLung-Study-A
Record Dates: First submitted 2022-12-09; First posted 2022-12-30 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Invasive Mechanical Ventilation
Keywords: Mechanical ventilation; ventilator-induced lung injury; ARDS; artificial intelligence
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Artificial Intelligence-based Decision support — Decision support to optimise invasive mechanical ventilation settings

SUMMARY:
Invasive mechanical ventilation is one of the most important and life-saving therapies in the intensive care unit (ICU). In most severe cases, extracorporeal lung support is initiated when mechanical ventilation is insufficient. However, mechanical ventilation is recognised as potentially harmful, because inappropriate mechanical ventilation settings in ICU patients are associated with organ damage, contributing to disease burden. Studies revealed that mechanical ventilation is often not provided adequately despite clear evidence and guidelines. Variables at the ventilator and extracorporeal lung support device can be set automatically using optimization functions and clinical recommendations, but the handling of experts may still deviate from those settings depending upon the clinical characteristics of individual patients. Artificial intelligence can be used to learn from those deviations as well as the patient's condition in an attempt to improve the combination of settings and accomplish lung support with reduced risk of damage.

ELIGIBILITY:
Inclusion Criteria:

• Subjects who are 18 years or older and receive invasive mechanical ventilation for > 4 hours

Exclusion Criteria:

• Patients receiving one-lung ventilation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Intensive care patients receiving invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 318542 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Relative time of same device settings of the health care provider and the IntelliLung algorithm | From date of intubation to date of extubation or date of discharge, which ever came first, assessed up to 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Wittenstein, MD, Principal Investigator — University Hospital Carl Gustav Carus at Technischen Universität Dresden, Germany
Locations (8):
- Cleveland Clinic Foundation, Cleveland, USA, Cleveland, Ohio, United States
- Germany (2):
  - University Hospital Carl Gustav Carus Dresden, Dresden
  - Institut Fur Angewandte Informatik (Infai) Ev, Leipzig
- Institut Mihajlo Pupin, Belgrade, Serbia
- Spain (3):
  - Better Care Sl, Sabadell
  - Fundacio Parc Tauli, Sabadell
  - Fundacion Publica Andaluza Progreso Y Salud, Seville
- Inselspital, Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No